CLINICAL TRIAL: NCT04178213
Title: First in Human Surgical Implantation of Single Piece ADAPT® Treated 3D ALR (Aortic Leaflet Repair), Feasibility and Clinical Safety Study
Brief Title: First in Human Feasibility Study With ADAPT 3D - ALR for Aortic Leaflet Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anteris Technologies Ltd. (Industry)
Collaborators: Factory CRO for Medical Devices B.V. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLRA-G012
Record Dates: First submitted 2019-11-19; First posted 2019-11-26 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Aortic Stenosis; Aortic Insufficiency
Keywords: ADAPT; aortic leaflet repair; aortic valve
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: prospective, non-randomised, single arm, single-centre First In Human clinical investigation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ADAPT 3D ALR (Experimental): Patients treated with ADAPT 3D ALR
  Interventions: Device: Implantation of ADAPT 3D ALR

INTERVENTIONS:
Device: Implantation of ADAPT 3D ALR — The operation is performed through a median sternotomy and with the hemodynamic support of standard cardiopulmonary bypass (CBP). diseased leaflets are excised meticulously. Calcifications at the level of the annulus will be removed just like in any other aortic valve replacement procedure. The annulus will be sized and the appropriate 3D single piece valve will be chosen. The implant technique will consist out of one running suture line at the level of the annulus, followed by fixation of the 3 commissural parts against the aortic wall. Valve competence and function will be assessed visually, and by TEE immediately coming of bypass.

SUMMARY:
This study will evaluate the safety and performance of the ADAPT 3D - ALR in adult patients requiring replacement of aortic valve. 15 patients in one site in Belgium will all be treated with ADAPT 3D - ALR.

DETAILED DESCRIPTION:
The purpose of this study is to conduct the initial clinical investigation of single piece ADAPT treated 3D - ALR (Aortic Leaflet Repair) to collect evidence on the device's safety and performance. The study is anticipated to confirm successful clinical safety and clinical performance with significant improvements in clinical hemodynamic performance.

The ADAPT® technology is used to process animal derived tissues to produce implantable tissue prosthetic devices that are compatible with the human body. This technology has been shown to produce reliable, biocompatible and versatile regenerative prosthetic devices capable of being used instead of synthetic products currently used in many soft tissue repair applications.

15 patients with aortic valve insufficiency or stenosis will be enrolled in this single arm single site study.

Follow-up will continue through to 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is older than 18 years of age and ≤ 85 years.
2. The subject's aortic annular measurements are ≥ 21 mm to < 27mm as confirmed on pre-op echo.
3. The subject is a candidate for Aortic Valve Replacement.
4. The subject has documented moderate or severe Aortic Stenosis and/or Aortic Insufficiency (defined as grade 2, 3 or 4).
5. The subject is willing and able to comply with specified follow-up requirements and evaluations, including transesophageal echocardiography (TEE) if there are inadequate images by transthoracic echocardiography (TTE) to assess the aortic valve.
6. Patient has signed the informed consent

Exclusion Criteria:

1. All patients who require emergency surgery (within 24 hours of a presentation to an emergency department) for any reason.
2. Subject with a pre-existing valve prosthesis in the aortic position.
3. Patients requiring repair of other cardiac valves will be excluded.
4. Subject with active endocarditis.
5. Heavily calcified aortic roots or "porcelain aortas".
6. Leukopenia with a WBC (white Blood Cells) of less than 3000.
7. Acute anaemia with a haemoglobin less than 8 g/dL.
8. Platelet count less than 100,000 platelets/microliter, and if less than 150,000 platelets/microliter, platelet reduction of >10,000 platelets/microliter per day over two consecutive days (Note: Where a platelet count is less than 150,000 platelets/microliter but greater than 100,000 platelets/microliter, platelet count testing is to be conducted over 2 consecutive days. If platelets are reducing over those two consecutive days, the rate of reduction in platelets must be less than 10,000 platelets/microliter per day, otherwise the participant must be excluded).
9. History of a defined bleeding diathesis or coagulopathy or the subject refuses blood transfusions.
10. Active infection requiring antibiotic therapy (if temporary illness, subjects may enroll 2-4 weeks after discontinuation of antibiotics).
11. Subjects in whom transesophageal echocardiography (TEE) is contraindicated.
12. Low EF < 50 %.
13. Life expectancy < 1 year, or severe comorbidities, such as cancer, dialysis, or severe COPD.
14. The subject is an illicit drug user, alcohol abuser, prisoner, institutionalised, or is unable to give informed consent.
15. The subject is pregnant or lactating (non-pregnancy to be confirmed by pregnancy test for all child bearing potential females).
16. Recent (within 6 months) cerebrovascular accident (CVA) or a transient ischemic attack (TIA).
17. Myocardial Infarction (MI) within one month of trial inclusion.
18. Currently participating in, or have been recently exited from (within 30 days of enrollment in this study), or plan to be enrolled in another clinical

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-03-26 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
mean pressure gradient (mmHg) across the valve (less than 20 mmHg) | 6 months following implantation
  Hemodynamic Performance Assessment
derived Effective Orifice Area (EOA) range > 0.9 cm2 (19mm valve) to > 1.6 cm2 (27mm valve) | 6 months following implantation
  Hemodynamic Performance Assessment
rate of thromboembolism | 6 months following implantation
  The adverse events consistent with the Objective Performance Criteria (OPC), for flexible heart valves will be compared to those rates defined as acceptable levels in the standard.
rate of valve thrombosis | 6 months following implantation
  The adverse events consistent with the Objective Performance Criteria (OPC), for flexible heart valves will be compared to those rates defined as acceptable levels in the standard.
rate of major paravalvular leak | 6 months following implantation
  The adverse events consistent with the Objective Performance Criteria (OPC), for flexible heart valves will be compared to those rates defined as acceptable levels in the standard.
rate of major hemorrhage | 6 months following implantation
  The adverse events consistent with the Objective Performance Criteria (OPC), for flexible heart valves will be compared to those rates defined as acceptable levels in the standard.
rate of endocarditis | 6 months following implantation
  The adverse events consistent with the Objective Performance Criteria (OPC), for flexible heart valves will be compared to those rates defined as acceptable levels in the standard.

SECONDARY OUTCOMES:
Rate of Atrial Fibrillation 6 months post procedure | 6 months post procedure
  New/post-operative atrial fibrillation - confirmed on ECG after closure till 6 months
number of days in ICU | 30 days post procedure
  Length of stay in the ICU post valve implantation defined as arrival time/date in hours and minutes to transfer to ward time/date in hours and minutes.
NYHA (New York Heart Association) class Improvement Assessment | 6 months post procedure
  Clinically significant improvement (one grade) in the New York Heart Association (NYHA) functional classification. 4 classes of disease: min value Class IV (cardiac disease resulting in inability to carry on any physical activity without discomfort); max value Class I (cardiac disease but without resulting limitations of physical activity)
number of days in hospital post procedure | 30 days post procedure
  Post procedure length of stay defined as the date and time in hours and minutes documented for arrival in the recovery unit to date and time in hours and minutes of discharge in hours and minutes.
hemoglobin assessment | 6 months post procedure
  Hemolysis screen measured by blood test
Alanine transaminase (ALT) | 6 months post procedure
  Hemolysis screen measured by blood test of liver enzyme
Aspartate transaminase (AST) | 6 months post procedure
  Hemolysis screen measured by blood test of liver enzyme
Rate of all-caused death | 6 months following implantation
  The rate will be compared to clinical outcomes for surgically implanted heart valves reported in the literature.
Rate of valve related death | 6 months following implantation
  The rate will be compared to clinical outcomes for surgically implanted heart valves reported in the literature.
Rate of valve-related reoperation | 6 months following implantation
  The rate will be compared to clinical outcomes for surgically implanted heart valves reported in the literature.
Rate of valve explant | 6 months following implantation
  The rate will be compared to clinical outcomes for surgically implanted heart valves reported in the literature.
Rate of hemorrhage | 6 months following implantation
  The rate will be compared to clinical outcomes for surgically implanted heart valves reported in the literature.
Rate of all-cause reoperation | 6 months following implantation
  The rate will be compared to clinical outcomes for surgically implanted heart valves reported in the literature.
Rate of Device deficiency | 6 months following implantation
  Device deficiency measured by echo

CONTACTS AND LOCATIONS:
Overall Officials: Bart Meuris, Prof. Dr., Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospital Leuven, Leuven, Belgium